CLINICAL TRIAL: NCT01766765
Title: Fast-track Surgery Recovery Program With Early Jejunostomy Nutrition Protocol Minimizes Time to Adjuvant Chemotherapy in Patients Undergoing Laparoscopic Gastrectomy for Gastric Cancer
Brief Title: Early Jejunostomy Nutrition Minimizes Time to Chemotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinling Hospital, China (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Qi Mao, Senior Resident, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EEN-001
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Gastric Cancer; Laparoscopic Surgery; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Jejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early jejunostomy nutrition (Experimental)
  Interventions: Procedure: Jejunostomy
- Early oral nutrition (Active Comparator)
  Interventions: Other: Early oral nutrition

INTERVENTIONS:
Procedure: Jejunostomy — Routine placement of jejunostomy tube following laparoscopic gastrectomy for gastric cancer. Immediately drip 37°C saline 20 ml/h and exchange to drip 37°C enteral nutrition fluid 20 ml/h at postoperative 6 h via jejunostomy tube
  Arms: Early jejunostomy nutrition
Other: Early oral nutrition — Free oral nutrition as tolerance allows on POD 1.
  Arms: Early oral nutrition

SUMMARY:
Adjuvant chemotherapy (AC) for gastric cancer is known to improve prognosis, and longer time to AC is associated with worse survival. However, most clinical trials mandate that AC is still to commence within 6 to 8 weeks after surgery consideration for malnutrition, postoperative complications and intolerance of AC. Placement of jejunostomy nutrition tube for enteral nutrition is a common component of these procedures, as a result of superior postoperative organ function, decreased infection rates, and a greater likelihood to complete AC with enteral nutritional support.

Fast-track surgery (FTS) recovery program focuses on enhancing recovery and reducing morbidity. Introduction of FTS concepts are safe, feasible, and can achieve shorter hospital stays and reduced costs. Early postoperative enteral nutrition combined with FTS results in reductions in total complications compared with traditional postoperative feeding practices and does not negatively affect outcomes. However, the benefit of jejunostomy nutrition tube routine placement and combination with FTS is still being debated. Besides, there remains some controversy over the optimal combination of nutrients and duration and timing and routes of feed administration.

The aim of this study was to determine whether FTS with early jejunostomy nutrition (EJN) following laparoscopic gastrectomy for gastric cancer improved postoperative recovery and minimizes time to AC when compared with FTS with early oral nutrition (EON).

ELIGIBILITY:
Inclusion Criteria:

* Primary gastric cancer
* R0 resection

Exclusion Criteria:

* Metastatic tumor
* Locally unresectable tumor
* Previous gastric/enteral resection
* Age under 18 years or over 70 years
* Preoperative complete parenteral or enteral nutrition
* Neo-adjuvant chemotherapy
* Severe malnutrition
* Lack of the patient's consent for the trial participation, jejunostomy tube insertion or epidural analgesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The time to the first adjuvant chemotherapy | 30 days after operation

SECONDARY OUTCOMES:
Overall morbidity rate of jejunostomy nutrition | 60 days after operation
Overall morbidity rate of early oral nutrition | 60 days after operation
Postoperative mortality rate | 60 days after operation
Time to tolerate EJN/EON | 30 days after operation
Time to full oral nutrition | 30 days after operation
Body composition | 10 days after operation
Energy metabolism | 10 days after operation
Postoperative hospital stay length | 60 days after operation
Rehospitalization rate | 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Qi Mao, MD/PhD, Principal Investigator — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] GASTRIC (Global Advanced/Adjuvant Stomach Tumor Research International Collaboration) Group; Paoletti X, Oba K, Burzykowski T, Michiels S, Ohashi Y, Pignon JP, Rougier P, Sakamoto J, Sargent D, Sasako M, Van Cutsem E, Buyse M. Benefit of adjuvant chemotherapy for resectable gastric cancer: a meta-analysis. JAMA. 2010 May 5;303(17):1729-37. doi: 10.1001/jama.2010.534. PMID 20442389
- [Background] Biagi JJ, Raphael MJ, Mackillop WJ, Kong W, King WD, Booth CM. Association between time to initiation of adjuvant chemotherapy and survival in colorectal cancer: a systematic review and meta-analysis. JAMA. 2011 Jun 8;305(22):2335-42. doi: 10.1001/jama.2011.749. PMID 21642686
- [Background] Osland E, Yunus RM, Khan S, Memon MA. Early versus traditional postoperative feeding in patients undergoing resectional gastrointestinal surgery: a meta-analysis. JPEN J Parenter Enteral Nutr. 2011 Jul;35(4):473-87. doi: 10.1177/0148607110385698. Epub 2011 May 31. PMID 21628607